CLINICAL TRIAL: NCT02232412
Title: Monitoring the Effect of Red Blood Cell Transfusion on Cerebral Oxygen Saturation With Near Infrared Spectroscopy (NIRS) in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr Dania Fischer, Dr. Dania Fischer, Johann Wolfgang Goethe University Hospital
Other Study IDs: NIRS-2014
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Effect of RBC Transfusions on Cerebral Oxygen Saturation
Keywords: Anemia; NIRS; Near Infrared Spectroscopy; RBC transfusion; critical ill; regional cerebral oxygen saturation; tissue oxygenation
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Critically ill patients are frequently transfused with red blood cell (RBC) units with the predominant intention to increase arterial oxygen content and thus oxygen delivery to the tissues.

To date, RBC transfusions have been proven effective in patients with profound anaemia or circulatory shock. However, the impact of the storage process and the so-called storage lesion on oxygen-carrying properties and, hence, the efficacy of RBC transfusion regarding tissue oxygenation are much debated at present. Alterations of RBC physiology have been comprehensively described ex vivo. Reduced deformability, increased adhesiveness and aggregability of stored RBC impair their rheological properties; anaerobic cellular metabolism with reduced contents of 2,3 bisphosphoglycerate and adenosine triphosphate (ATP) increases oxygen affinity and impairs oxygen release to the tissues.

This study aims to monitor the effect RBC transfusion has on the regional cerebral oxygen saturation (rSO2) of critically ill patients. rSO2 will be measured indirectly, using near infrared spectroscopy (NIRS) . Patients will be monitored once it looms that they might require RBC transfusion. The monitoring is continued for the time of transfusion and the hours afterwards.

ELIGIBILITY:
Inclusion Criteria:

* expected requirement of RBC transfusion
* 18 yrs and older

Exclusion Criteria:

* severe traumatic brain injury (Glasgow coma scale < 9), subarachnoid hemorrhage (Hunt and Hess scale ≥ 3) or intracranial hemorrhage
* cerebral ischaemia
* active bleeding
* patients necessitating ongoing resuscitation
* deficient signal of rSO2 impeding its proper valuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients requiring haemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
regional cerebral oxygen saturation (rSO2) | 24-48 hours
  Regional cerebral oxygen saturation (rSO2) will be measured before, during and after RBC transfusion. As the decision to transfuse is multifactorial and the condition of critically ill patients often instable, time frames before, during and after transfusion may vary.

CONTACTS AND LOCATIONS:
Overall Officials: Kai D Zacharowski, MD, PhD, FRCA, Study Director — University Hospital Frankfurt, Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy; Patrick Meybohm, MD, Study Chair — University Hospital Frankfurt, Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy; Dania P Fischer, MD, Principal Investigator — University Hospital Frankfurt, Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany